CLINICAL TRIAL: NCT06871644
Title: CD7CAR-T Cell Therapy As a Single-Arm, Open-Label, Single-Center Investigator-Initiated Early-Stage Clinical Study
Brief Title: Clinical Study of CD7 CAR-T Cells for Relapsed/refractory Autoimmune Diseases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-007-8
Record Dates: First submitted 2025-02-27; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Systemic Sclerosis - 2013 ACR/EULAR Classification Criteria

STUDY DESIGN:
Intervention Model Description: CD7 CAR-T cell therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- T cell injection targeting CD7 chimeric antigen receptor (Experimental): CD7 CAR-T cell therapy Subjects meeting the inclusion/exclusion criteria will be entered into the 0.25×108, 1×108, and 2×108 CAR-T groups in sequential order, and will be administered once
  Interventions: Biological: T cell injection targeting CD7 chimeric antigen receptor

INTERVENTIONS:
Biological: T cell injection targeting CD7 chimeric antigen receptor — Subjects who sign the informed consent form and meet the inclusion/exclusion criteria will be entered into the 0.25×108, 1×108 and 2×108 CAR-T groups, in order of priority, and will be administered 1 dose of

SUMMARY:
The primary objective was to evaluate the safety of CD7 CAR-T cells for the treatment of subjects with relapsed/refractory AID. CD7 CAR-T cells were infused in a single infusion in subjects who were screened after signing an informed consent form and undergoing single nucleus cell collection and pretreatment, and blood was collected before and after the infusion for pharmacokinetic, pharmacodynamic, immunogenicity, and safety evaluations.

DETAILED DESCRIPTION:
Subjects who meet the inclusion/exclusion criteria will be entered into 3 groups in sequential order for a single dose. The dose-escalation study utilizes a "3+3" design, i.e., 3-6 subjects in each group will complete a single dose.

After the last subject in each dose group completes a dose-limiting toxicity (DLT) assessment window of 28 days after the single dose, enrollment in the next dose group can begin.

When 1 DLT occurs in 3 subjects in a dose group, 3 additional subjects are required in the same dose group (up to 6 subjects in that dose group have completed DLT assessment): if no DLT occurs in the 3 additional subjects, continue the dose escalation; if 1 of the 3 additional subjects develops a DLT, stop the dose escalation; if >1 of the 3 additional subjects DLT occurs, the dose escalation is stopped and a one-dose reduction is required to continue enrolling 3 more subjects for DLT assessment.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed relapsing/refractory systemic sclerosis that has failed treatment with at least two immunosuppressive and/or biologic agents.

Bone marrow and coagulation function, liver and kidney function, cardiopulmonary function are satisfied No serious mental disorders

Exclusion Criteria:

- Malignancy other than AID disease within 5 years prior to screening Hepatitis B surface antigen (HBsAg) positive, AIDS, syphilis and other virus positive persons Severe heart disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-18 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
adverse events | About 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
（Cmax） | About 1 year
  Maximum concentration of CD7 CAR-T cells expanded in peripheral blood after drug administration
（Tmax） | About 1 year
  Time to maximum concentration
AUC0-28d | About 28 days
  Area under the curve at 28 days
AUC0-90d | About 90 days
  Area under the curve at 90 days
Disease remission rate | About 90 days
  Rate of decline from baseline in the American College of Rheumatology Composite Response Index (ACR-CRISS)

CONTACTS AND LOCATIONS:
Overall Officials: zhu chen, doctor, Principal Investigator — The First Hospital Affiliated to the University of Science and Technology of China
Locations (1):
- PersonGen.Anke Cellular Therapeutice Co. Ltd, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes
Research details